CLINICAL TRIAL: NCT04050982
Title: Feasibility Study to Improve Atrial Fibrillation Outcomes Using a Digital Application for Cardiovascular Risk Reduction: Precursor to a Multicenter Randomized Trial
Brief Title: Feasibility Study to Improve AF Outcomes Using a Digital Application for CV Risk Reduction
Acronym: AFCARE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Acquisition of digital messaging company and decision made to withdraw study support
Sponsor: Stanford University (Other)
Collaborators: American Heart Association (Other); PatientBond (Industry)
Responsible Party: Principal Investigator, Paul Wang, Director, Stanford Electrophysiology and Arrhythmia Service, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB# 48183
Record Dates: First submitted 2019-08-07; First posted 2019-08-09 (Actual); Results first posted 2023-09-22 (Actual); Last update posted 2023-09-22 (Actual); Status verified 2023-08

CONDITIONS: Atrial Fibrillation
Keywords: Text Messaging; Patient Education; Psychometric
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Intervention Model Description: Randomized control trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (3):
- Pilot Testing (Experimental): Patients interface with the digital application, providing feedback on usability and satisfaction.
  Interventions: Device: AF CARE
- AF CARE plus Usual Care (Active Comparator): Patients will interface with the digital application.
  Interventions: Device: AF CARE; Behavioral: Usual Care
- Usual Care then AF Care (Active Comparator): After a 6 month period of usual care only, patients will interface with the digital application.
  Interventions: Behavioral: Usual Care

INTERVENTIONS:
Device: AF CARE — Patients will receive personalized messages twice weekly that will include behavior recommendations for CVRF reduction and AF education based on the initially entered psychographic profile and data entered.
  Arms: AF CARE plus Usual Care; Pilot Testing
Behavioral: Usual Care — Participants will be given recommendations for CVRF reduction based on their initial American Heart Association Life Simple 7 (LS7) assessment and will be provided educational materials and be wait listed for digital app 3 months later
  Arms: AF CARE plus Usual Care; Usual Care then AF Care

SUMMARY:
The pilot portion of this study is to determine the feasibility of utilizing AF CARE to provide lifestyle modification support to patients with atrial fibrillation (AF).

The prospective, RCT portion of this study compare cardiovascular risk factors (CVRF), AF knowledge, AF Symptom Severity and Burden, and QOL between and within the wait list group and the AF CARE group at baseline, 3, 6, and 12 months.

ELIGIBILITY:
Inclusion Criteria:

1. BMI > 28 kg/m2 AND one additional CVRF using LS7
2. Access and willingness to engage in digital technology
3. Has a valid email address and a cell phone number
4. Able to ambulate
5. Able to speak/read English

Exclusion Criteria:

1. Class III/IV heart failure
2. MI or cardiac surgery in prior 3 months
3. Severe renal/hepatic disease
4. Active malignancy
5. Current/recent (within 6 months) enrollment in weight loss program

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2023-01-26 (Actual); Study Completion 2023-01-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Linda Ottoboni, PhD, Principal Investigator — Clinician and research scientist
Locations (1):
- Stanford Health Care, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Pilot Testing: Patients interface with the AF CARE digital platform, providing feedback on usability and satisfaction.
- AF CARE Plus Usual Care: Patients interface with the AF CARE digital platform and receive usual care.
- Usual Care Then AF Care: After a 6 month period of usual care only, patients will interface with the AF CARE digital platform.
Period: Overall Study
Arm/Group | Pilot Testing | AF CARE Plus Usual Care | Usual Care Then AF Care
Started | 9 | 2 | 0
Interfaced With AF CARE Digital Platform | 7 | 1 | 0
Completed | 7 | 1 | 0
Not Completed | 2 | 1 | 0
Not completed — Did not meet eligibility criteria | 0 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0
Not completed — Unable to enroll on platform | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pilot Testing | AF CARE Plus Usual Care | Total
Number analyzed (Participants) | 9 | 2 | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 1 | 6
  >=65 years | 4 | 1 | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 2 | 7
  Male | 4 | 0 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 9 | 2 | 11
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 6 | 2 | 8
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 9 | 2 | 11

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Text Messages That Were Reviewed
Time Frame: Baseline through month 6
Population: Data for this outcome measure were collected only in the Pilot Testing group. Only participants who interfaced with the AF CARE platform are included.
Measure: Mean (Full Range); unit: percentage of texts
Arm/Group | Pilot Testing
Number analyzed (Participants) | 7
percentage of texts | 29.2 [0 to 60.0]

2. Primary Outcome: Percentage of Emails Opened and Clicked Through
Description: Percentage of emails opened, and of those opened, the percentage of emails clicked through
Time Frame: Baseline through month 6
Population: as for outcome 1
Measure: Mean (Full Range); unit: percentage of emails
Arm/Group | Pilot Testing
Number analyzed (Participants) | 7
percentage of emails
  Emails opened | 72.2 [19 to 97]
  Emails clicked through | 74.3 [36 to 100]

3. Primary Outcome: Cardiovascular Risk Factor Score
Description: The American Heart Association Life Simple 7 (LS7) is a calculated score using lab values, biometric measurements, and patient dietary responses. Score range: 0 to 10; 0 = most risk, 10 = least risk
Time Frame: Baseline, month 3, month 6, and month 12
Population: Data for this outcome measure were collected only in the AF CARE plus Usual Care group. Only participants who interfaced with the AF CARE platform are included.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | AF CARE Plus Usual Care
Number analyzed (Participants) | 1
score on a scale
  baseline | 6.5 (0)
  month 3 | 8 (0)
  month 6 | 6.5 (0)
  month 12 | 7 (0)

4. Secondary Outcome: Change From Baseline in Knowledge Related to Atrial Fibrillation
Description: AF knowledge assessed with the Jessa AF Knowledge Score calculated from a 16 question self- reported questionnaire with a scoring range from 0-16, 16 indicating greater knowledge.
Time Frame: Baseline, month 3, month 6, and month 12
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | AF CARE Plus Usual Care
Number analyzed (Participants) | 1
score on a scale
  baseline | 12 (0)
  month 3 | 11 (0)
  month 6 | 15 (0)
  month 12 | 15 (0)

5. Secondary Outcome: Change From Baseline in AF Quality of Life Score
Description: Quality of Life assessed using a patient completed questionnaire, Atrial Fibrillation Effect on Quality of Life Questionnaire (AFEQT). The AFEQT score is a combined score of 21 items; overall score range is 21 to 100, with a higher score representing greater QOL.
Time Frame: Baseline, month 3, month 6, and month 12
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | AF CARE Plus Usual Care
Number analyzed (Participants) | 1
score on a scale
  baseline | 82 (0)
  month 3 | 65 (0)
  month 6 | 67 (0)
  month 12 | 51 (0)

6. Secondary Outcome: Change From Baseline in AF Symptom Severity
Description: AF symptom severity assessed with the Atrial Fibrillation Symptoms Severity Scale (AFSS). The AFSS is a patient self-reported questionnaire that contains 21 questions, with 7 questions that provide calculated scores for AF symptom severity (0-35) with higher scores representing greater severity.
Time Frame: Baseline, month 3, month 6, and month 12
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | AF CARE Plus Usual Care
Number analyzed (Participants) | 1
score on a scale
  baseline | 0 (0)
  month 3 | 15 (0)
  month 6 | 21 (0)
  month 12 | 23 (0)

7. Secondary Outcome: Change From Baseline in AF Symptom Burden
Description: AF symptom burden assessed with the Atrial Fibrillation Symptom Severity Scale. The AFSS is a patient self-reported questionnaire that contains 21 questions that provides calculated scores for AF Burden, calculated in the following manner; AF Burden = AF frequency + AF duration + AF severity. Each of the 3 measures contribute equally to the AF burden score, and each measure ranges from 1-10 to yield Total AF Burden scores ranging from 3-30. Higher scores indicate greater AF burden.
Time Frame: Baseline, month 3, month 6, and month 12
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | AF CARE Plus Usual Care
Number analyzed (Participants) | 1
score on a scale
  baseline | 2 (0)
  month 3 | 16 (0)
  month 6 | 19 (0)
  month 12 | 22 (0)

ADVERSE EVENTS:
Time Frame: Up to 12 months
Arm/Group | Pilot Testing | AF CARE Plus Usual Care
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/2
Other Adverse Events (participants affected / at risk) | 0/9 | 0/2

LIMITATIONS AND CAVEATS:
The study did not meet its planned enrollment size, and did not achieve statistical power.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-05-17): https://cdn.clinicaltrials.gov/large-docs/82/NCT04050982/Prot_SAP_000.pdf